CLINICAL TRIAL: NCT01355185
Title: Seed Movement in Prostate Brachytherapy Implants: Clinical Measurement and Dosimetric Consequences
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Canadian Association of Radiation Oncology (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: 25750
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Prostate Cancer
Keywords: Seed movement; implants; prostate brachytherapy; localized
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
There are substantial uncertainties with contemporary seed placement techniques in prostate brachytherapy, particularly with the impact of seed movement after an implant due to edema and migration of seeds in the prostate and peri-prostatic tissues. This study will accrue 20 patients undergoing prostate brachytherapy implants and perform serial CT and MRI scans at specified intervals (pre-operatively, day 0, day 3, day 10 and day 28) to characterize these phenomena.

DETAILED DESCRIPTION:
Prostate brachytherapy is an effective treatment option for men with localized prostate cancer with excellent cure rates and a favorable toxicity profile. Having a more detailed understanding of seed movement after an implant will provide clinicians with details about the clinical impact of these phenomena on implants and provide the detailed understanding of these phenomena that are necessary for more sophisticated brachytherapy implants that are envisioned in the future.

ELIGIBILITY:
Inclusion Criteria:

* treated with prostate brachytherapy
* low risk or intermediate risk prostate cancer
* ambulatory
* stable medical condition
* 18 years of age or older
* capable of informed consent

Exclusion Criteria:

* no use of any hormonal therapy
* unable to have MRI scans (ie. presence of metallic foreign object, aneurysm clip, cardiac pacemaker, internal wires, implanted pump, implanted cardiac device, claustrophobia, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen at an academic institution (tertiary centre ...Cross Cancer Institute) for consideration of prostate brachytherapy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-08; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nawaid Usmani, MD, FRCPC, Principal Investigator — University of Alberta; Ronald Sloboda, PhD, Principal Investigator — University of Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Sloboda RS, Usmani N, Pedersen J, Murtha A, Pervez N, Yee D. Time course of prostatic edema post permanent seed implant determined by magnetic resonance imaging. Brachytherapy. 2010 Oct-Dec;9(4):354-61. doi: 10.1016/j.brachy.2009.09.008. Epub 2010 Jan 29. PMID 20116344